CLINICAL TRIAL: NCT06702540
Title: Bio-reconfigurable Differential Impedance Electronic Platform for High Sensitivity Multiplex Detection of Viral Respiratory Pathogens
Brief Title: Bio-reconfigurable Electronic Platform for Multiplex Detection of Viral Respiratory Pathogens
Acronym: BIOPLEX
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Politecnico di Milano (Other); Consiglio Nazionale delle Ricerche, Italy (Unknown)
Responsible Party: Principal Investigator, Nicola Clementi, Associate professor of Microbiology and Virology, IRCCS San Raffaele
Other Study IDs: BIOPLEX 2022EJL28B; 2022EJL28B (Other Grant/Funding Number: Ministero dell'Università e della Ricerca (MUR))
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: COVID 19
Keywords: COVID-19; SARS-CoV-2; Biosensor chip
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Analyses performed on plasma samples already stored with nasopharyngeal swabs during the first pandemic COVID-19 waves according to the San Raffaele institutional COVID-19 clinical-biological biobank (COVID-BioB, NCT04318366) procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Positive for respiratory viruses: 79 retrospective samples tested positive for respiratory viruses
  Interventions: Device: Biosensor chip
- Negative to respiratory viruses: 79 retrospective samples tested negative to respiratory viruses
  Interventions: Device: Biosensor chip

INTERVENTIONS:
Device: Biosensor chip — An electronic platform measuring the impedance variation between microelectrodes is used upon capturing the target biomolecule by a selective bioprobe previously grafted over the biosensor surface. The required sensitivity will be achieved by operating the biosensor in lock-in mode, which ensures the highest resolution in tracking amplitude and phase variations of impedance signals.

SUMMARY:
This project focuses on developing a cutting-edge electronic biosensor platform for highly sensitive and specific detection of target biomolecules, with initial applications targeting SARS-CoV-2 detection. The system operates on impedance measurement between microelectrodes, utilizing lock-in mode for unparalleled resolution (1 ppm). Enhanced signal detection is achieved via functionalized polystyrene microbeads that amplify impedance changes, building on prior success in Dengue virus antibody detection.

Key innovations include Differential Impedance Sensing across multiple channels for real-time comparative analysis of various targets, and a biosensor chip modified with DMA-based functional polymers for optimal probe immobilization and target interaction. The biosensor integrates with a pre-existing microfluidic system and supports whole-virus detection using DNA-labelled antibodies against SARS-CoV-2 spike protein, coupled with complementary oligonucleotide-functionalized beads. This strategy is complemented by antigen-specific detection for practical applications such as point-of-care testing in pharmacies.

The project includes a retrospective study analyzing anonymized respiratory and plasma samples from a COVID-19 biobank to validate the platform's sensitivity in detecting viral particles. These efforts aim to advance diagnostic technologies for respiratory infections with a focus on safety, scalability, and versatility.

DETAILED DESCRIPTION:
The project stands on the development of an electronic platform performing the measurement of the impedance variation between microelectrodes upon the capture of the target biomolecule by a selective bioprobe previously grafted over the biosensor surface. The required sensitivity will be achieved by operating the biosensor in lock-in mode, which ensures the highest resolution in tracking amplitude and phase variations of impedance signals (1 ppm has been demonstrated by POLIMI on other applications). To enhance the electronic signal, polystyrene microbeads, properly functionalized with oligonucleotides or antibodies, are used to link the target and increase the impedance variation as demonstrated by proponents in the successful detection of antibodies against Dengue virus. To address multiple sensing sites in parallel on the same biosensor chip, allowing real-time comparative analysis on different targets from the same biological sample for augmented detection sensitivity and control, a custom-made electronic platform will be developed to perform Differential Impedance Sensing (i.e., direct comparison between the target sensor and a reference) on multiple channels. The biosensor chip, made of borosilicate with gold microelectrodes, features a specific modification of its surface with functional polymers (a family of N,N-dimethylacrylamide -DMA-based polymers) developed by CNR that form a nanometric hydrophilic film on the chip surface. The functional groups of these copolymers allow the covalent immobilization of the probe preserving its active structure, proper spatial distance, orientation and density, favoring the interaction with the target. The biosensor chip will be integrated into the microfluidic system already available in the group.

SARS-CoV-2 will be targeted with challenging strategies. First, we plan to capture the entire virus in solution using DNA-labelled antibodies directed against the SARS-CoV-2 spike protein.

The sensor area, spotted with oligonucleotide probes complementary to the DNA sequence linked to the antibody, will interact with the DNA-labelled antibodies which have decorated the entire surface of the virus. To increase the impedance variation of the platform polystyrene beads will be used: in particular, they will be modified with the oligonucleotide complementary to that linked to the antibody which have captured the virus. This entire-virus detection methodology, combining the DNA-directed capture of the antigens together with a high sensitivity platform for Differential Impedance Sensing, is absolutely new and expected to be successful based upon the results already achieved by the proponents in the detection of the antibodies in the human blood of persons infected by Dengue virus. In parallel, we intend to extend the use of the electronic platform also to the detection of viral antigens, i.e. Spike protein S or nucleocapside protein N. The use of antigens for the diagnosis of the infection instead of the entire virus, may lead to important practical dropouts as it does not necessitate any particular safety requirement, thus allowing the test to be performed in any location, in particular pharmacies or medical clinics similarly to standard antigenic lateral flow tests.

This is a retrospective monocenter study to test respiratory samples to evaluate the analytical sensitivity of the platform being developed in the project PRIN Prot. 2022EJL28B. The samples are completed anonymized and the samples analyses are performed in order to check the ability of the device to reveal the presence of viral particles in biological matrix such as respiratory samples or, when necessary for set up of instruments, plasma randomized and anonymized samples. No patients or use of clinical data will be involved for the study, but only used the samples stored in the San Raffaele institutional COVID-19 clinical-biological biobank (COVID-BioB, NCT04318366). The samples used for the study were collected during the period 19/03/2020 - 31/05/2024.

ELIGIBILITY:
Inclusion Criteria:

* Samples tested for respiratory viruses, stored at the San Raffaele institutional COVID-19 clinical-biological biobank (COVID-BioB, NCT04318366).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: No patients or use of clinical data will be involved for the study, but only used the samples stored in the San Raffaele institutional COVID-19 clinical-biological biobank (COVID-BioB, NCT04318366). The samples used for the study were collected during the period 19/03/2020 - 31/05/2024.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Validation of the biosensor platform with nasopharyngeal swabs | 12 months
  Real-time impedance measurement in randomized respiratory samples to detect respiratory viruses

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu W, Liu L, Kou G, Zheng Y, Ding Y, Ni W, Wang Q, Tan L, Wu W, Tang S, Xiong Z, Zheng S. Evaluation of Nucleocapsid and Spike Protein-Based Enzyme-Linked Immunosorbent Assays for Detecting Antibodies against SARS-CoV-2. J Clin Microbiol. 2020 May 26;58(6):e00461-20. doi: 10.1128/JCM.00461-20. Print 2020 May 26. PMID 32229605
- [Background] Seo G, Lee G, Kim MJ, Baek SH, Choi M, Ku KB, Lee CS, Jun S, Park D, Kim HG, Kim SJ, Lee JO, Kim BT, Park EC, Kim SI. Rapid Detection of COVID-19 Causative Virus (SARS-CoV-2) in Human Nasopharyngeal Swab Specimens Using Field-Effect Transistor-Based Biosensor. ACS Nano. 2020 Apr 28;14(4):5135-5142. doi: 10.1021/acsnano.0c02823. Epub 2020 Apr 20. PMID 32293168
- [Background] Sola L, Damin F, Gagni P, Consonni R, Chiari M. Synthesis of Clickable Coating Polymers by Postpolymerization Modification: Applications in Microarray Technology. Langmuir. 2016 Oct 11;32(40):10284-10295. doi: 10.1021/acs.langmuir.6b02816. Epub 2016 Sep 29. PMID 27632284
- [Background] Piedimonte P, Sola L, Cretich M, Gori A, Chiari M, Marchisio E, Borga P, Bertacco R, Melloni A, Ferrari G, Sampietro M. Differential Impedance Sensing platform for high selectivity antibody detection down to few counts: A case study on Dengue Virus. Biosens Bioelectron. 2022 Apr 15;202:113996. doi: 10.1016/j.bios.2022.113996. Epub 2022 Jan 15. PMID 35091373
- [Background] F. Morichetti et al., "Non-Invasive On-Chip Light Observation by Contactless Waveguide Conductivity Monitoring," in IEEE Journal of Selected Topics in Quantum Electronics, vol. 20, no. 4, pp. 292-301, July-Aug. 2014, Art no. 8201710, doi: 10.1109/JSTQE.2014.2300046.
- [Background] Ciccarella, Pietro et al. "Multichannel 65 zF rms Resolution CMOS Monolithic Capacitive Sensor for Counting Single Micrometer-Sized Airborne Particles on Chip." IEEE Journal of Solid-State Circuits 51 (2016): 2545-2553.